CLINICAL TRIAL: NCT00091741
Title: A Phase I Pilot Study to Evaluate Safety and Efficacy of Etanercept (Enbrel) on the Response Rate of HIV-infected Subjects Who Are in Virologic Failure and Who Have Failed to Respond to Standard Antiretroviral Therapy
Brief Title: Safety and Efficacy Study of Etanercept (Enbrel) on the Response Rate of HIV-infected Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Advanced Biotherapy, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 03-365
Record Dates: First submitted 2004-09-16; First posted 2004-09-20 (Estimated); Last update posted 2009-07-22 (Estimated); Status verified 2004-09

CONDITIONS: HIV Infection
Keywords: HIV; Treatment Experienced; Complementary Therapies
MeSH Terms: conditions — HIV Infections | interventions — Etanercept

INTERVENTIONS:
Drug: Etanercept (Enbrel)

SUMMARY:
The purpose of conducting this already-FDA approved Phase I clinical trial is to evaluate the safety and efficacy of etanercept (Enbrel) on the response rate in HIV-infected subjects who have failed to respond to conventional antiretroviral (HAART) therapy and for whom no alternative therapy exists. The greatest challenge faced by HIV-treating clinicians today is the management of virologic failure and metabolic complications of anti-HIV treatment. Treatment failure can occur because of non-compliance, drug discontinuation, lack of drug potency, inadequate drug plasma concentration or drug resistance. Of these, drug resistance remains the single most important reason for virological failure and rapidly limits treatment options.

DETAILED DESCRIPTION:
I. Background and Rationale:

The greatest challenge faced by HIV-treating clinicians today is the management of virologic failure and metabolic complications of anti-HIV treatment. Treatment failure can occur because of non-compliance, drug discontinuation, lack of drug potency, inadequate drug plasma concentration or drug resistance. Of these, drug resistance remains the single most important reason for virological failure and rapidly limits treatment options. Virus resistance to all three major antiretroviral drug classes is now being reported even in primary seroconverters. Although highly-active antiretroviral (ARV) therapy (HAART) has led to a sharp decline in AIDS-related morbidity and mortality, treatment failure is a common, significant problem and as many as 50% of patients have detectable plasma HIV RNA despite being on combination ARV therapy. Salvage therapy is the term commonly used to define the approach taken when previous anti-HIV treatments fail to achieve desired goals, which include: 1) undetectable viral load; 2) CD4 cell levels below 200 cells/mm3; and, 3) the prevention of HIV disease progression. It is one of the most difficult situations to face as a patient, and one of the most problematic challenges for health-care providers. Although this state of treatment failure is sometimes euphemistically referred to as "management of treatment-experienced patients," many HIV positive patients, having already exhausted the benefits of at least a few drug combinations, think of their next regimen as salvage or "rescue" therapy. Some physicians argue that due to cross-resistance among different drugs within the same class, people with HIV infection have only one good shot at treating it, and that any treatment regimen beyond the first is therefore salvage therapy. Others see salvage therapy as literally the end of the line--when an individual's HIV has developed extensive resistance to all currently available treatments. But most providers consider salvage therapy to be somewhere in between these extremes. Data on salvage therapy mostly comes from anecdotal reports and retrospective cohort studies. With a paucity of clinical trial data, clinicians are often forced to prescribe unproven regimens based on what is anticipated about cross-resistance and drug interactions. It is important, therefore, that new agents and new approaches continue to be developed as an increasing number of patients in practice have exhausted all treatment options.

The rationale of this study is based upon the existing literature which indicates that many of the manifestations and subsequent clinical deterioration of HIV-infected individuals are related to the immune dysfunction seen in HIV disease, many of which are caused by the overproduction of proinflammatory cytokines, most notable of which is the excessive production of TNF-α. It is further postulated that removal of this TNF-α by a commercially available TNF-α-binding medication [ENBREL (etanercept)] may provide therapeutic benefit for HIV-infected patients who have failed to respond to standard antiretroviral therapy.

II. Goal and Objectives:

The purpose of the project is to assess the safety profile and efficacy of a soluble p75 tumor necrosis factor (TNF) receptor: Fc fusion protein (Enbrel; Amgen, (etanercept) Thousand Oaks, CA) [i.e. anti TNF-α] on the response rate of "salvage patients" who are in virologic failure and who have failed to respond to standard antiretroviral therapy.

The protocol will evaluate:

1. Changes in CD4 T-cell enumeration, viral load, and soluble immune activation markers in HIV-infected patients from baseline to week 24 following treatment with anti-TNF-α.
2. Safety and tolerability of anti-TNF-α with respect to treatment-limiting symptoms and laboratory adverse events through week 24.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years.
* Confirmed diagnosis of HIV-1 infection, as documented by any licensed ELISA test kit, and confirmed by Western blot at any time prior to study entry, HIV-1 culture, HIV-1 antigen, plasma HIV-1 RNA.
* Prior antiretroviral therapy, defined as: Receipt of at least two separate protease inhibitor (PI)-containing regimens (minimum 12 weeks) which was changed because of virological failure (per subject or physician history) or detectable plasma HIV-1 RNA AND A minimum of 1 year total prior antiretroviral experience.
* A CD4 count of > 200.
* Signed a written informed consent prior to initiation of any study related procedures.
* All subjects should continue taking the same antiretroviral regimen between the screening and entry visits.

Exclusion Criteria:

* History or suspicion of active tuberculosis or a prior history of being treated for tuberculosis.
* Documented history of sepsis.
* Known hypersensitivity to ENBREL or any of its components.
* Patients on concomitant immunosuppressive therapy, e.g., steroids, cyclosporine, etc.
* Any condition which may interfere with the trial, including the patient's mental ability to follow protocol instructions.
* Patients with heart failure or a history of congestive heart failure.
* Renal insufficiency (creatinine >2.5 mg/dL)
* Women of child bearing potential who are not willing to avoid pregnancy for the duration of the study and 3 months thereafter.
* Inability or unwillingness to take appropriate prophylaxis for opportunistic infections (i.e., PCP toxoplasmosis, etc.)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Study Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Georgetown University Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] De SK, Devadas K, Notkins AL. Elevated levels of tumor necrosis factor alpha (TNF-alpha) in human immunodeficiency virus type 1-transgenic mice: prevention of death by antibody to TNF-alpha. J Virol. 2002 Nov;76(22):11710-4. doi: 10.1128/jvi.76.22.11710-11714.2002. PMID 12388730
- [Background] Zagury D, Burny A, Gallo RC. Toward a new generation of vaccines: the anti-cytokine therapeutic vaccines. Proc Natl Acad Sci U S A. 2001 Jul 3;98(14):8024-9. doi: 10.1073/pnas.141224798. PMID 11438746